CLINICAL TRIAL: NCT06153732
Title: The Foot Posture and Falling Risk in Older People
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Bahar Anaforoglu Külünkoglu (Other)
Responsible Party: Sponsor-Investigator, Bahar Anaforoglu Külünkoglu, Associate Professor, Ankara Yildirim Beyazıt University
Organization: Ankara Yildirim Beyazıt University (Other)
Other Study IDs: AnkaraYBU
Record Dates: First submitted 2023-11-23; First posted 2023-12-01 (Actual); Last update posted 2023-12-08 (Actual); Status verified 2023-12

CONDITIONS: Aged
Keywords: Falls; Aged; Foot

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This research will be conducted to examine the relationship between the foot postures and fall risks of elderly individuals living in nursing homes, to identify the factors that most affect the risk of falling, and to inform healthcare professionals working on this subject.

Factors that may increase the risk of falling will be determined from the biomechanical changes that occur in the foot with age. In addition, the results we obtain will contribute to the database to be created in the future to identify factors affecting the risk of falling.

DETAILED DESCRIPTION:
The aim of this study is to examine the relationship between foot postures and fall risks of elderly individuals living in nursing homes, to identify the factors that most affect the risk of falling and to inform healthcare professionals on this subject.

Participants included in the research will be grouped in three ways according to their gender, disease status and whether they use medication or not. The disease conditions of the participants will be handled in two ways: direct and indirect disease groups due to falls.

The researchers will evaluate the cognitive status of the participants with the Standardized Mini Mental State Test, balance and fall risks of the participants with the One Leg Standing Test and the 8 Step Up and Go Test and foot postures of the participants with the Foot Posture Index.

A power analysis was conducted to determine the number of participants required for the research. According to the power analysis result; It was found that the minimum number of participants required to be included in the study for one-way analysis of variance with an effect size of 0.3, α= 0.05, and 85% power was 126.

Ethics committee approval for the research was received by the researchers from Ankara Yıldırım Beyazıt University Health Sciences Ethics Committee on 05.01.2020 with research number 2020-600. Later, the researchers made the necessary applications to conduct this study in Karadeniz Ereğli İzmirlioğlu Nursing Home, affiliated with the Zonguldak Provincial Directorate of Family and Social Services.

However, due to the Covid-19 pandemic that affected the whole world, permission approval for the study for the Karadeniz Ereğli İzmirlioğlu Nursing Home was given to the researchers by the Zonguldak Provincial Directorate of Family and Social Services on January 21, 2022. In the preliminary examination conducted by the researchers, it was determined that the number of people required to be included in the study could not be reached from only one nursing home.

For this reason, the researchers again applied to Ankara Yıldırım Beyazıt University Health Sciences Ethics Committee with the request to add new nursing homes to the study.

In order to expand the scope of the research and conduct it in Zonguldak Center and Çaycuma Nursing Homes, a new ethics committee permission was obtained with the decision of Ankara Yıldırım Beyazıt University Health Sciences Ethics Committee dated 09.06.22 and numbered 10/960.

Later, the researchers made the necessary applications to conduct this study in Zonguldak Center and Çaycuma Nursing Homes affiliated with the Zonguldak Provincial Directorate of Family and Social Services.

Permission approval to conduct the study in Zonguldak Center and Çaycuma Nursing Homes was given to the researchers by the Zonguldak Provincial Directorate of Family and Social Services on August 11, 2022. Participants who meet the inclusion and exclusion criteria, aged 65 and over, living in Zonguldak Center and Çaycuma Nursing Home, will be included in the research.

ELIGIBILITY:
Inclusion Criteria:

* 65 years and older
* Scoring 24 and above from the Mini Mental State Test
* Completing the 8 step up and go test in the Senior Fitness Test Protocol

Exclusion Criteria:

* Those who need the use of auxiliary tools in performing daily life activities,
* Those who are in the recovery period of an acute disease,
* Cancer patients known to be life-threatening,
* Cardiovascular problem (previous congestive heart failure, transient ischemic attacks),
* Parkinson's disease,
* Stroke history in the last 6 months
* Progressive neuromuscular disease,
* Acute inner ear inflammation and severe hearing loss,
* Those who have lost their eyesight enough to be unable to read the test protocol and see the movements in the test,
* Those who have a fall story in the last year,
* Those who are in a structured exercise program more than three times a week (not physically active),
* Those with chronic orthopedic diseases

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Zonguldak Center, Çaycuma and Kdz, affiliated to the Zonguldak Provincial Directorate of Family and Social Services, participated in the study. Volunteer elderly individuals living in Ereğli İzmirlioğlu Nursing Homes who meet the inclusion criteria will participate in the study.An application will be made to Zonguldak Provincial Directorate of Family and Social Services to conduct this study and the necessary permissions will be obtained. The work will begin after receiving permission approval from the relevant units.
Sampling Method: Non-Probability Sample
Enrollment: 126 (Estimated)
Dates: Start 2023-01-02 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Mini Mental State Test | Baseline
  For Individuals; A questionnaire consisting of 2 questions about recording memory, 1 about attention and calculation, 1 about remembering, 6 questions about language, 10 questions about orientation and a maximum total score of 30 will be applied. From the MMDT scores; 28-30 range; high normal, 24-27 range indicates low cognitive function, and 0-23 range indicates impaired cognitive status.

SECONDARY OUTCOMES:
Eight Step Up and Go Test included in the Senior Fitness Test: | Baseline
  It is performed at a distance of 2.44 cm, using a chair with a straight back and no armrest with a seat height of 43.18 cm, a meter, a cone, a stopwatch with an accuracy of 1/10 second. When the individual gets up from the chair with the start command while sitting position, the stopwatch is started with the command. The individual is asked to turn around the cue point at a distance of 2.44 cm as quickly as possible, but without running, and reach the chair again.

OTHER OUTCOMES:
Stand on One Foot Test: | Baseline
  For balance evaluation, a one-leg standing test will be performed on the right and left sides.
  The participant is asked to alternately stand on the right and left foot, with the other foot bent at knee level for 30 seconds.
  After the participant takes the desired position, measurements will be made 3 times, both with eyes open and with eyes closed, for a maximum of 30 seconds, and the average value will be calculated in seconds.
  The test will be terminated if the participant's upper foot touches the ground, jumps with his foot on the ground, or opens his eyes.
Foot Posture Index | Baseline
  The test score is calculated by assigning values between -2 and +2 to the 6 criteria on the foot and summing the scores from all criteria. A test score of 0 indicates that the foot is in a neutral position. A positive test score indicates standing pronation. A negative test score indicates standing supination.

CONTACTS AND LOCATIONS:
Overall Officials: Bahar ANAFOROGLU KULUNKOGLU, Assoc. Prof., Principal Investigator — Ankara Yildirim Beyazıt University
Locations (1):
- Zonguldak Center, Kdz. Ereğli İzmirlioğlu and Çaycuma Nursing Homes, Zonguldak, Center, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No